CLINICAL TRIAL: NCT05930691
Title: Evaluation of the Association Between the Optic Nerve Sheath Diameter and Extracorporeal Life Support Time During Cardiac Surgery in Newborn
Brief Title: Optic Nerve Sheath Diameter and the Duration of Extracorporeal Life Support During Newborn Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Aydın Mermer, Vice Director, Head of Anesthesiology, Principal Investigator, Clinical Speicialist, Konya City Hospital
Other Study IDs: 2023/4253
Record Dates: First submitted 2023-06-02; First posted 2023-07-05 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Extracorporeal Life Support
Keywords: Pediatric Cardiovascular surgery; Optic Nerve Sheath diameter; intracranial pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Optic nerve sheath diameter measurement — Prediction of intracranial pressure by using Ultrasonography on optic nerve sheath diameter.

SUMMARY:
Mortality rates for newborns with congenital heart disease (CHD) have dramatically decreased thanks to surgical methods and medical treatment improvements. Up to 70% of patients may have post- Extracorporeal life support (ECLS) cerebral dysfunction, which can result in long-term cognitive and motor impairment, first showing as brain edema and higher intracranial pressure (ICP). Optic Nerve Sheath Diameter (ONSD) is a non-invasive method of measuring Intracranial Pressure (ICP). The Primary Aim of this study is to identify the correlation between ONSD and ECLS time in newborns who get ECLS.

DETAILED DESCRIPTION:
INTRODUCTION Mortality rates for newborns with congenital heart disease (CHD) have dramatically decreased thanks to surgical methods and medical treatment improvements. As a result, more emphasis is being put on reducing neonatal cardiac surgery morbidity.

Extracorporeal life support (ECLS) is increasingly being given to children, particularly for cardiac causes, according to the Pediatric Extracorporeal Life Support Organization Registry's global report. However, up to 70% of patients may have post-ECLS cerebral dysfunction, which can result in long-term cognitive and motor impairment, first showing as brain edema and higher intracranial pressure (ICP). In addition, pediatric patients may have trouble being diagnosed with acute elevations in IİCP since the signs and symptoms are sometimes unclear.

The gold standard for measuring intracranial pressure (ICP) still involves invasive intracranial devices. In addition, ICP monitors have the potential to cause complications, including bleeding in 1.1-5.8% of cases, malfunction, in 6.3-40% of cases, or infection in 0-15% of cases, with a noticeable higher risk of bacterial colonization after five days.

The optic nerve sheath surrounds the Optic Nerve (ON) and covers the optic subarachnoid space, which is connected to the intracranial subarachnoid space area. Changes in intracranial pressure are thus straightly transferred to the optic nerve sheath. Therefore, Optic Nerve Sheath Diameter (ONSD) is a non-invasive method of measuring Intracranial Pressure (ICP).

Longer ECLS periods and aortic cross-clamp times have been linked to more frequent CT detection of cerebral edema, according to prior investigationsAccording to prior investigations, long ECLS periods, and aortic cross-clamp times have been linked to more frequent CT (computer tomography) detection of cerebral edema. However, there is currently no information on the relationship between these time points and the ONSD determined by ultrasound.

The Primary Aim of this study was to identify the correlation between ONSD and ECLS time in newborns who get ECLS. Specifically, we tested the primary hypothesis that more ECLS time means more ONSD valuable over the perioperative period. Our secondary aim was to investigate the relationship between ONSD and aortic cross-clamp time and operation time and also, operation time and preoperative and intraoperative perioperative ONSD variation for the ECLS period.

ELIGIBILITY:
Inclusion Criteria:

* ASA III or IV status newborn;
* Have surgery for transposition of great arteries (TGA).

Exclusion Criteria:

* All off-pump cardiac surgery;
* Recent history of cerebrovascular accident or intracranial hypertension due to any cause;
* History of increased ICP;
* Ophthalmological diseases capable of affecting optic nerve diameters.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will occur newborns and will have cardiac surgery because of the surgery for transposition of great arteries (TGA). We worked on sample size analyses and found that it should be 22 patients at least to reach our actual power.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Correlation between optic nerve sheath diameter and extra corperal support life time. | Basal; the 15. minutes after aort cross clamp; the time of removing cross clamp; End of the operation.
  The Primary outcome of this study will be identifing ONSD in ECLS time in newborns.

SECONDARY OUTCOMES:
Staticticaly meaningful between Cross clamp time and optic nerve sheath diameter | Basal; the 15. minutes after aort cross clamp; the time of removing cross clamp; End of the operation.
  Our secondary outcome will be ONSD in aortic cross-clamp time.
Staticticaly meaningful between operation time and optic nerve sheath diameter | Basal; the 15. minutes after aort cross clamp; the time of removing cross clamp; End of the operation.
  Our secondary outcome will be ONSD in operation time.
Perioperative ONSD variation for the ECLS period. | Basal; the 15. minutes after aort cross clamp; the time of removing cross clamp; End of the operation.
  Our secondary outcome will be ONSD variation for the ECLS period.

CONTACTS AND LOCATIONS:
Overall Officials: Aydın Mermer, MD, Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided